CLINICAL TRIAL: NCT00110292
Title: An RCT of a Low-Intensity Intervention to Reduce Delay
Brief Title: Preventing Learning Problems in Young Children: A Public Health and Physician-Based Outreach
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: R01HD040388 (NIH)
Record Dates: First submitted 2005-05-05; First posted 2005-05-06 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-05

CONDITIONS: Developmental Disabilities; Language Development Disorders
Keywords: Public health; Primary care; Parenting education; Child rearing; Parenting newsletters; Child development; Language delay
MeSH Terms: conditions — Developmental Disabilities; Language Development Disorders

INTERVENTIONS:
Behavioral: Age-specific parenting newsletters and developmental toys
Behavioral: Parent-completed Ages & Stages Questionnaires
Behavioral: Clinic-based distribution of children's books

SUMMARY:
This study will evaluate a program to prevent learning problems in children. The program is an inexpensive public health outreach program designed for families living in poverty and is administered through pediatricians' offices and clinics.

DETAILED DESCRIPTION:
This study will assess the effectiveness of a low-intensity, low-cost, preventive intervention to reduce developmental delay and learning problems in young children. The goal is to improve home caregiving environment factors that are often suboptimal in families living in poverty; these families are often subject to social, economic, and medical risk factors. The intervention is based on a public health/primary care partnership and combines mailed parent-completed Ages & Stages Questionnaires (ASQ), a monthly mailed age-paced parenting newsletter (Building Blocks) and corresponding developmental toys (BB), and a Reach Out and Read (ROR) physician-based distribution of children's books.

Families of 4- to 7-month-old children attending a participating pediatric clinic will be randomized to either an ASQ/BB+ROR group, an ROR-only group, or a no intervention control group. Outcomes measures will be obtained at 15, 24, 36, and 48 months of age and include measures of the home environment, parenting and parent-child interaction, child language and mental development measures, and rates of referral to Early Intervention programs. Baseline and ongoing demographic information and psychosocial and biological risk factors will also be gathered to see how they relate to child and family outcomes and to determine whether certain subgroups of families are more likely to benefit from the intervention than others.

ELIGIBILITY:
Inclusion Criteria

* Attend participating pediatric clinic (serving poor, largely black, and Hispanic communities)
* Family with child 4 to 7 months of age at enrollment
* English- or Spanish-speaking

Exclusion Criteria

* Developmental delay
* Eligible for Early Intervention program

Ages: 4 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600
Dates: Start 2002-03; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Overall Officials: Harris S. Huberman, MD, Principal Investigator — Medical & Health Research Association of NYC, Inc.
Locations (2):
- United States (2):
  - Montefiore Comprehensive Health Care Center, The Bronx, New York
  - North Central Bronx Hospital Pediatric Clinic, The Bronx, New York